CLINICAL TRIAL: NCT01206140
Title: Randomized, Phase II Trial of AZD6244 Alone and AZD6244 Plus Temsirolimus for Soft-Tissue Sarcomas
Brief Title: Selumetinib With or Without Temsirolimus in Treating Patients With Metastatic, Recurrent, or Locally Advanced Soft Tissue Sarcoma That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: National Comprehensive Cancer Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02532; NCI-2011-02532 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000685408; CHNMC-PHII-95; NCCN-T06; PHII-95 (Other: City of Hope Comprehensive Cancer Center); 8412 (Other: CTEP); N01CM00038 (NIH); P30CA033572 (NIH)
Record Dates: First submitted 2010-09-18; First posted 2010-09-21 (Estimated); Results first posted 2015-10-05 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2015-01

CONDITIONS: Recurrent Adult Soft Tissue Sarcoma; Stage III Adult Soft Tissue Sarcoma; Stage IV Adult Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — AZD 6244; temsirolimus; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (selumetinib and temsirolimus) (Experimental): Patients receive selumetinib PO twice daily on days 1-28 and temsirolimus IV over 30-60 minutes on days 1, 8, 15, and 22.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Selumetinib; Drug: Temsirolimus
- Arm II (selumetinib) (Experimental): Patients receive selumetinib as in arm I. Patients who experience disease progression may cross over to arm I.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Selumetinib

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Selumetinib — Given PO
  Other Names: ARRY-142886; AZD6244; MEK Inhibitor AZD6244
Drug: Temsirolimus — Given IV
  Other Names: CCI-779; CCI-779 Rapamycin Analog; Cell Cycle Inhibitor 779; Rapamycin Analog; Rapamycin Analog CCI-779; Torisel
  Arms: Arm I (selumetinib and temsirolimus)

SUMMARY:
This randomized phase II trial is studying how well giving selumetinib together with or without temsirolimus works in treating patients with metastatic, recurrent, or locally advanced soft tissue sarcoma that cannot be removed by surgery. Selumetinib and temsirolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known whether giving selumetinib together with temsirolimus is more effective than giving selumetinib alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Compare the progression-free survival of the MEK inhibitor, AZD6244 (selumetinib) alone, and the combination of AZD6244 and a mammalian target of rapamycin inhibitor (mTORi), temsirolimus (CCI-779) in patients with recurrent metastatic or recurrent locally unresectable soft-tissue sarcomas.

SECONDARY OBJECTIVES:

I. Determine the rates of apoptosis, autophagy, and proliferation with AZD6244 alone, and in combination with temsirolimus by immunohistochemistry in tumor and surrogate skin tissue biopsies. (exploratory) II. Assess the activation status of protein kinase B (Akt), 5E-BP1, eukaryotic translation initiation factor 4 gamma, 1 (eIF-4G), and ribosomal protein S6 kinase (S6K) in tumor biopsy samples and surrogate skin tissue biopsy samples.(exploratory) III. Assess inhibition of activated mitogen-activated protein kinase 1/2 (ERK1/2) in stimulated peripheral blood mononuclear cells. (exploratory) IV. Assess response by Choi criteria. V. Compare the response rate and 4-month progression-free survival (PFS) rate in patients treated with these regimens.

VI. Compare the response rate, 4-month PFS rate and toxicity of AZD6244 alone and in combination with temsirolimus.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive selumetinib orally (PO) twice daily on days 1-28 and temsirolimus intravenously (IV) over 30-60 minutes on days 1, 8, 15, and 22.

ARM II: Patients receive selumetinib as in arm I. Patients who experience disease progression may cross over to arm I.

In both arms, courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have had histologic verification of soft-tissue sarcoma at original diagnosis (GIST subtype is eligible)
* Patients must have metastatic (de novo or recurrent) or locally advanced, unresectable disease; patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques or as >= 10 mm with spiral CT scan
* ECOG 0-2 (Karnofsky >= 50%)
* Patients may have received 0-2 prior cytotoxic chemotherapeutic regimens for metastatic or recurrent disease (single-agent or combination chemotherapies)
* Estimated life expectancy > 12 weeks
* Peripheral absolute neutrophil count (ANC) >= 1000/uL
* Platelet count >= 100,000/uL (transfusion independent)
* Hemoglobin >= 8.0 gm/dL (may receive RBC transfusions)
* Creatinine =< 1.5 x upper institutional limits of normal, or calculated creatinine clearance >= 45mL/min, based on the Cockcroft-Gault formula
* Bilirubin (sum of conjugated + unconjugated) =< 1.5 x upper limit of normal (ULN) for age
* SGPT (ALT) =< 5 x upper limit of normal (ULN) for age
* No evidence of dyspnea at rest, no exercise intolerance
* Pulse oximetry > 94% if there is clinical indication for determination
* For women: must be surgically sterile, postmenopausal, or compliant with a medically approved contraceptive regimen (for example, intrauterine device [IUD], birth control pills, or barrier device) during and until 4 weeks after the last dose of study treatment; must have a negative serum or urine pregnancy test within 7 days before study enrollment, and must not be breast-feeding; should a woman become pregnant or suspect she is pregnant while she or her partner participating in this study, the patient should inform her treating physician immediately; for men: must be surgically sterile or compliant with a contraceptive regimen during and for 16 weeks after the treatment period; please note that the AZD6244 manufacturer recommends that adequate contraception for male patients should be used for 16 weeks post-last dose due to sperm life cycle
* All patients must sign a written informed consent

Exclusion Criteria:

* Patients with pediatric-type sarcomas (Ewing's or primitive neuroectodermal tumor, rhabdomyosarcoma, and desmoplastic small round cell tumor)
* Concomitant Medications

  * Growth factor(s): growth factors that support platelet or white cell number or function must not have been administered within the past 7 days
  * Steroids: patients with CNS tumors who have not been on a stable or decreasing dose of dexamethasone for the past 7 days
  * Investigational Drugs: patients who are currently receiving another investigational drug
  * Anti-cancer Agents: patients who are currently receiving other anti-cancer agents; at least 3 weeks must have elapsed since prior chemotherapy or radiation (6 weeks for mitomycin-C and nitrosureas)
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to AZD6244
* Previous MEK inhibitor use
* Patients with QTc interval > 450 msecs or other factors that increase the risk of QT prolongation or arrhythmic events (e.g., heart failure, hypokalemia, family history of long QT interval syndrome); this may be determined by either Bazett's correction (QTc =QT/RR0.5) or Friderica's correction (QTc = QT/RR0.33); QTc exclusion > 450 msec requires calculation according to both formulas
* Patients unable to swallow the AZD6244 capsules are ineligible
* Refractory nausea and vomiting, chronic gastrointestinal diseases (e.g., inflammatory bowel disease), or significant bowel resection that would preclude adequate absorption
* Uncontrolled intercurrent illness including, but not limited to, uncontrolled, ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because the effects of AZD6244 on the developing human fetus at the recommended therapeutic dose are unknown; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother, breastfeeding should be discontinued if the mother is treated with AZD6244
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with AZD6244; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study
* Prior cardiac history of uncontrolled hypertension, New York Heart Association (NYHA) Classification >= class II, current or prior cardiomyopathy, baseline LVEF < 50%, ongoing atrial fibrillation, recent myocardial infarction or unstable ischemic heart disease
* Concomitant Strong CYP1A2 or CYP3A4 inducers and/or inhibitors; prior treatment with an mTOR inhibitor for recurrent soft-tissue sarcoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2010-10; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Warren Chow, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (8):
- United States (8):
  - Tower Cancer Research Foundation, Beverly Hills, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - University of California Davis Phase 2 Consortium, Sacramento, California
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Selumetinib): Patients receive 75 mg selumetinib as in arm II. Patients who experience disease progression may cross over to arm II.
  Laboratory Biomarker Analysis: Correlative studies
  Selumetinib: Given PO
- Arm II (Selumetinib and Temsirolimus): Patients receive selumetinib 75 mg PO twice daily on days 1-28 and temsirolimus 25 mg IV over 30-60 minutes on days 1, 8, 15, and 22.
  Laboratory Biomarker Analysis: Correlative studies
  Selumetinib: Given PO
  Temsirolimus: Given IV
Period: Overall Study
Arm/Group | Arm I (Selumetinib) | Arm II (Selumetinib and Temsirolimus)
Started | 35 | 35
Completed | 34 | 35
Not Completed | 1 | 0
Not completed — Deemed ineligible due to incorrect diag. | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Selumetinib) | Arm II (Selumetinib and Temsirolimus) | Total
Number analyzed (Participants) | 34 | 35 | 69
Age, Continuous [Median (Full Range); unit: years] | 56 [34 to 84] | 56 [20 to 83] | 56 [20 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 25 | 42
  Male | 17 | 10 | 27
Region of Enrollment [Number; unit: participants]
  United States | 34 | 35 | 69

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progression-free survival was estimated using the product-limit method of Kaplan and Meier. Progression wasl evaluated in this study using the Response Evaluation Criteria in Solid Tumors (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions, or death.
Time Frame: Until disease progression or death, up to 4.5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Selumetinib) | Arm II (Selumetinib and Temsirolimus)
Number analyzed (Participants) | 34 | 35
months | 1.8 [0.5 to 1.8] | 3.7 [1.6 to 9.3]

2. Secondary Outcome: Number of Participants With Objective Response
Description: Response evaluated using the Choi criteria. CR - disappearance of all lesions and no new lesions; PR - a decrease in size (the sum of longest diameters of target lesions as defined in RECIST) of 10% or more or a decrease in tumor density (HU) of 15% or more on CT and no new lesions and no obvious progression of nonmeasurable disease; SD - does not meet the criteria for CR, PR, or PD and no symptomatic deterioration attributed to tumor progression; PD - an increase in tumor size of 10% or more and does not meet criteria of PR by tumor density (HU) on CT or new lesions or new intratumoral nodules or increase in the size of the existing intratumoral nodules. Objective response = CR+PR.
Time Frame: Evaluated for response after every two cycles, up to 4.5 years.
Measure: Number; unit: participants
Arm/Group | Arm I (Selumetinib) | Arm II (Selumetinib and Temsirolimus)
Number analyzed (Participants) | 34 | 35
participants | 5 | 4

3. Secondary Outcome: 4 -Month Progression-free Survival Rate.
Description: Progression-free survival rate was calculated using the survival distribution function, and 95% confidence limits were calculated using the log-log transformation. Progression was defined using the Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions, or death.
Time Frame: Four months
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Arm I (Selumetinib) | Arm II (Selumetinib and Temsirolimus)
Number analyzed (Participants) | 34 | 35
percent of participants | 24 [9 to 40] | 24 [9 to 39]

ADVERSE EVENTS:
Time Frame: Adverse events collected over a period of 28 months
Description: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Arm/Group | Arm I (Selumetinib) | Arm II (Selumetinib and Temsirolimus)
Serious Adverse Events (participants affected / at risk) | 23/34 | 18/35
Other Adverse Events (participants affected / at risk) | 33/34 | 35/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Selumetinib) (N=34) | Arm II (Selumetinib and Temsirolimus) (N=35)
Anemia (Blood and lymphatic system disorders) | 3 (5) | 1 (1)
Aortic valve disease (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Volume overload (Cardiac disorders) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 4 (5) | 1 (1)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (3) | 0 (0)
Duodenal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal obstruction (Gastrointestinal disorders) | 2 (3) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (2)
Oral pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2)
Chills (General disorders) | 1 (1) | 0 (0)
Edema face (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 3 (3) | 0 (0)
Fever (General disorders) | 2 (4) | 1 (1)
Injection site reaction (General disorders) | 2 (2) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
vaginal mucositis (General disorders) | 0 (0) | 1 (1)
Biliary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Bladder infection (Infections and infestations) | 0 (0) | 1 (1)
Bronchial infection (Infections and infestations) | 1 (1) | 0 (0)
Catheter related infection (Infections and infestations) | 1 (2) | 1 (1)
Device related infection (Infections and infestations) | 2 (2) | 1 (1)
Endocarditis infective (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 3 (3) | 1 (1)
Paronychia (Infections and infestations) | 3 (4) | 1 (1)
Penile infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (3) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Unknown source but positive blood cultur (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Viral gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
left groin area (Infections and infestations) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Alkaline phosphatase increased (Investigations) | 2 (3) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 1 (1)
Ejection fraction decreased (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 4 (5) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Weight gain (Investigations) | 1 (1) | 0 (0)
Weight loss (Investigations) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 4 (5) | 4 (4)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (5) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (4) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Progressive disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 2 (2) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Genital edema (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Spinal cord compression (Surgical and medical procedures) | 1 (1) | 0 (0)
T5 Laminectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 6 (18) | 1 (1)
Hypotension (Vascular disorders) | 3 (3) | 0 (0)
Lymphedema (Vascular disorders) | 2 (2) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Selumetinib) (N=34) | Arm II (Selumetinib and Temsirolimus) (N=35)
Anemia (Blood and lymphatic system disorders) | 25 (98) | 27 (73)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 1 (2)
Murmer (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 2 (2) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 2 (2)
Sinus bradycardia (Cardiac disorders) | 1 (3) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 7 (14) | 5 (5)
pedal edema (Cardiac disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 2 (3)
Middle ear inflammation (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Cushingoid (Endocrine disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Blepharitis (Eye disorders) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 2 (2) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (2) | 3 (3)
Dry eye (Eye disorders) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 1 (1) | 3 (6)
Floaters (Eye disorders) | 2 (2) | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 1 (1)
Scleral disorder (Eye disorders) | 0 (0) | 1 (1)
disconjugate gaze (Eye disorders) | 1 (1) | 0 (0)
drainage (Eye disorders) | 1 (1) | 0 (0)
left eye conjunctival hemorrhage (Eye disorders) | 0 (0) | 1 (1)
right eye conjunctival hemorrhage (Eye disorders) | 0 (0) | 1 (1)
swollen left eye (Eye disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 6 (6) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 12 (18) | 4 (4)
Bloating (Gastrointestinal disorders) | 3 (3) | 2 (4)
Colonic hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 17 (35) | 11 (14)
Dark Stool (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 18 (31) | 15 (22)
Dry mouth (Gastrointestinal disorders) | 6 (8) | 6 (7)
Dyspepsia (Gastrointestinal disorders) | 3 (4) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 1 (2)
Esophageal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Esophageal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Esophageal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 5 (7) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4 (4) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gum Abscess (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 15 (30) | 24 (46)
Nausea (Gastrointestinal disorders) | 22 (51) | 13 (18)
Oral pain (Gastrointestinal disorders) | 2 (2) | 8 (9)
Rectal fistula (Gastrointestinal disorders) | 0 (0) | 1 (2)
Rectal hemorrhage (Gastrointestinal disorders) | 3 (3) | 0 (0)
Rectal mucositis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 2 (3) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 18 (40) | 12 (15)
mucoid diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 9 (12) | 8 (16)
Edema face (General disorders) | 6 (12) | 11 (12)
Edema limbs (General disorders) | 17 (52) | 14 (24)
Edema trunk (General disorders) | 1 (2) | 0 (0)
Fatigue (General disorders) | 28 (93) | 18 (35)
Fever (General disorders) | 8 (15) | 8 (11)
Flu like symptoms (General disorders) | 2 (4) | 2 (3)
Gait disturbance (General disorders) | 3 (5) | 1 (2)
Infusion related reaction (General disorders) | 1 (1) | 1 (1)
Injection site reaction (General disorders) | 1 (1) | 2 (2)
Localized edema (General disorders) | 1 (1) | 1 (2)
Malaise (General disorders) | 1 (1) | 0 (0)
Night Sweats (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 7 (8) | 0 (0)
Pain (General disorders) | 5 (15) | 2 (5)
dry nose (General disorders) | 1 (1) | 0 (0)
night sweats (General disorders) | 0 (0) | 1 (1)
stent replaced - obstructed by tumor (Hepatobiliary disorders) | 1 (1) | 0 (0)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (4)
Catheter related infection (Infections and infestations) | 0 (0) | 1 (1)
Eye infection (Infections and infestations) | 0 (0) | 2 (3)
Mucosal infection (Infections and infestations) | 1 (1) | 1 (1)
Papulopustular rash (Infections and infestations) | 2 (2) | 0 (0)
Paronychia (Infections and infestations) | 2 (10) | 1 (1)
Penile infection (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (2)
R big toe infection (Infections and infestations) | 1 (2) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 4 (9) | 5 (8)
Thrush (Infections and infestations) | 0 (0) | 2 (2)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1)
infected necrotic tumor (Infections and infestations) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (3)
Fracture (Injury, poisoning and procedural complications) | 1 (6) | 0 (0)
Activated partial thromboplastin time pr (Investigations) | 2 (2) | 2 (4)
Alanine aminotransferase increased (Investigations) | 11 (24) | 10 (13)
Alkaline phosphatase increased (Investigations) | 9 (27) | 14 (29)
Aspartate aminotransferase increased (Investigations) | 19 (53) | 18 (28)
Blood bilirubin increased (Investigations) | 3 (4) | 1 (1)
CD4 lymphocytes decreased (Investigations) | 1 (1) | 3 (5)
CPK increased (Investigations) | 1 (1) | 0 (0)
Cholesterol high (Investigations) | 10 (48) | 13 (29)
Creatinine increased (Investigations) | 4 (5) | 4 (11)
INR increased (Investigations) | 2 (7) | 5 (7)
Lipase increased (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 6 (12) | 14 (38)
Lymphocyte count increased (Investigations) | 0 (0) | 1 (2)
Neutrophil count decreased (Investigations) | 11 (25) | 14 (44)
Platelet count decreased (Investigations) | 15 (42) | 24 (49)
QTc prolonged (Investigations) | 0 (0) | 1 (1)
Weight gain (Investigations) | 2 (7) | 0 (0)
Weight loss (Investigations) | 5 (11) | 3 (7)
White blood cell decreased (Investigations) | 12 (42) | 14 (43)
alanine aminotransferase decreased (Investigations) | 1 (1) | 0 (0)
eosinophilia (Investigations) | 0 (0) | 1 (1)
ionized calcium (Investigations) | 0 (0) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 14 (34) | 15 (21)
Chloride increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 6 (16) | 13 (27)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (4) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 11 (36) | 13 (26)
Hypoalbuminemia (Metabolism and nutrition disorders) | 20 (37) | 18 (37)
Hypocalcemia (Metabolism and nutrition disorders) | 7 (14) | 11 (16)
Hypoglycemia (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 8 (14) | 13 (28)
Hypomagnesemia (Metabolism and nutrition disorders) | 4 (8) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 11 (34) | 9 (13)
Hypophosphatemia (Metabolism and nutrition disorders) | 7 (11) | 3 (7)
Increased LDH (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
LDH increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 7 (50) | 2 (4)
increased LDH (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (7) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (14) | 6 (8)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 4 (16) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 4 (6) | 0 (0)
Generalized body aches (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 4 (6) | 4 (4)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 (5) | 0 (0)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (11) | 2 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (5) | 2 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 (34) | 9 (13)
Pelvic soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
muscle cramps (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
muscle spasm, left hip (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
shoulder pain (L) w/ cough (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
twitching (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (36) | 2 (5)
Ataxia (Nervous system disorders) | 1 (1) | 1 (1)
Concentration impairment (Nervous system disorders) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 4 (16) | 4 (8)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 6 (17) | 6 (9)
Facial muscle weakness (Nervous system disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 7 (9) | 4 (4)
L facial palsy (Nervous system disorders) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 6 (6) | 1 (1)
Memory impairment (Nervous system disorders) | 3 (3) | 1 (1)
Myelitis (Nervous system disorders) | 0 (0) | 1 (2)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 4 (6) | 2 (2)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 1 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 2 (3)
Phantom pain (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 1 (1)
Radiculitis (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 3 (5) | 3 (3)
Spasticity (Nervous system disorders) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 2 (3) | 1 (1)
Anxiety (Psychiatric disorders) | 5 (8) | 5 (5)
Confusion (Psychiatric disorders) | 1 (1) | 2 (2)
Depression (Psychiatric disorders) | 6 (12) | 4 (7)
Insomnia (Psychiatric disorders) | 11 (21) | 6 (8)
Libido decreased (Psychiatric disorders) | 3 (11) | 2 (3)
Lucid per physical exam (Psychiatric disorders) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 0 (0) | 2 (3)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 3 (3)
Nocturia (Renal and urinary disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 5 (5) | 2 (2)
Renal calculi (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Urine discoloration (Renal and urinary disorders) | 3 (3) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (8) | 1 (1)
Genital edema (Reproductive system and breast disorders) | 2 (9) | 0 (0)
Irregular menstruation (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 3 (11) | 1 (1)
Penile pain (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal dryness (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal mucositis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chest Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 14 (41) | 7 (9)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 15 (39) | 9 (16)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (8) | 7 (7)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (15) | 3 (3)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 (7) | 2 (2)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (4)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (26) | 6 (11)
Dry skin (Skin and subcutaneous tissue disorders) | 6 (23) | 6 (11)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Nail discoloration (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Nail loss (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Nail ridging (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Palmar-plantar erythrodysesthesia syndro (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Periorbital edema (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (5) | 9 (19)
Rash acneiform (Skin and subcutaneous tissue disorders) | 22 (67) | 17 (40)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 (8) | 8 (12)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 2 (10) | 1 (1)
Telangiectasia (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
burning in armpits (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
cut on palm (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
folliculitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
ingrown toe nail (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
pin point rash/non red/dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
pin point rash/non-red/dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
redness and liquid in stump area (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
small fissures on finger pads (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (2)
Hot flashes (Vascular disorders) | 2 (3) | 0 (0)
Hypertension (Vascular disorders) | 19 (81) | 12 (33)
Hypotension (Vascular disorders) | 3 (3) | 1 (1)
Lymphedema (Vascular disorders) | 1 (10) | 4 (6)
Thromboembolic event (Vascular disorders) | 2 (6) | 3 (3)
venous stasis changes, legs (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less